CLINICAL TRIAL: NCT00139594
Title: A 52-week, Open-label Extension Study to Evaluate the Safety and Tolerability of Licarbazepine in the Treatment of Manic Episodes of Bipolar I Disorder
Brief Title: Open Label Extension Study of Licarbazepine in the Treatment of Manic Episodes of Bipolar I Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC477D2303E1
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder, manic episode/treatment/licarbazepine
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

ARMS (1):
- licarbazepine (Experimental)
  Interventions: Drug: licarbazepine

INTERVENTIONS:
Drug: licarbazepine

SUMMARY:
This extension study is designed to assess the long-tem tolerability and safety of licarbazepine in patients who completed the 6-week double-blind study CLIC477D2303.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent provided prior to participation in the extension study
* successful completion of study CLIC477D2303
* cooperation and willingness to comply with all study requirements

Exclusion Criteria:

* premature discontinuation from study CLIC477D2303
* failure to comply with study CLIC477D2303

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of treatment with licarbazepine over 52 weeks.
with respect to the rates of adverse events and serious adverse events, as well as changes in laboratory values, ECGs and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (13):
  - Investigational site, La Palma, California
  - Novartis Investigational Site, Kansas City, Kansas
  - Novartis Investigational Site, Shreveport, Louisiana
  - Novartis Investigational Site, Somerville, Massachusetts
  - Novartis Investigational Site, Farmington Hills, Michigan
  - Novartis Investigational Site, Staten Island, New York
  - Novartis Investigational Site, Madison, Tennessee
  - Novartis Investigational Site, Bellaire, Texas
  - Novartis Investigational Site, Dallas, Texas
  - Novartis Investigational Site, Verdun, Texas
  - Novartis Investigational Site, Bellevue, Washington
  - Novartis Investigational Site, Kirkland, Washington
  - Novartis Investigational site, West Allis, Wisconsin
- Novartis Investigational Site, Vienna, Austria
- Canada (5):
  - Novartis Investigational Site, Greater Sudbury
  - Novartis Investigational Site, Kelowna
  - Novartis Investigational Site, London
  - Novartis Investigational Site, Montreal
  - Novartis Investigator Site, Vancouver
- Colombia (3):
  - Novartis Investigational Site, Bogotá
  - Novartis Investigational Site, Medellín
  - Novartis Investigational Site, Pareira
- Czechia (3):
  - Novartis Investigational Site, Brno
  - Novartis Investigational Site, Hradec Králové
  - Novartis Investigational Site, Prague
- Germany (6):
  - Novartis Investigational Site, Berlin
  - Novartis Investigational Site, Bochum
  - Novartis Investigational Site, Dresden
  - Novartis Investigational Site, Ingolstadt
  - Novartis Investigational Site, Mannheim
  - Novartis Investigational Site, Würzburg
- Novartis Investigational Site, Guatemala City, Guatemala
- Novartis Investigational Site, Lima, Peru
- Russia (2):
  - Novartis Investigational Site, Moscow
  - Novartis Investigational Site, Yaroslavl
- Slovakia (2):
  - Novartis Investigational Site, Bojnice
  - Novartis Investigational Site, Michalovce
- Novartis Investigational Site, Durban, South Africa
- Ukraine (5):
  - Novartis Investigational Site, Dnipro
  - Novartis Investigational Site, Kiev
  - Novartis Investigational Site, Luhansk
  - Novartis Investigational Site, Odesa
  - Novartis Investigational Site, Simferopol
- Novartis Investigational Site, Caracas, Venezuela